CLINICAL TRIAL: NCT06230250
Title: Unilateral Secondary Breast Reconstruction Using a Muscle-sparing Pedicled Dorsal Flap in Patients With a History of Total Mastectomy for Breast Cancer Single-centre Observational Study
Brief Title: Unilateral Secondary Breast Reconstruction Using a Muscle-sparing Pedicled Dorsal Flap After Breast Cancer
Acronym: RMSU-LDPEM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BREC23.0196 - RMSU-LDPEM
Record Dates: First submitted 2024-01-08; First posted 2024-01-30 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-01

CONDITIONS: Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The use of pedicled dorsal flaps sparing the latissimus dorsi muscle (TDAP and MSLD flap) is a well-described reconstruction method in breast reconstruction after breast cancer. However, little data exists regarding patient satisfaction after this surgery. The main objective of this study was to evaluate patient satisfaction after unilateral total secondary breast reconstruction using a TDAP or MSLD flap.

ELIGIBILITY:
Inclusion Criteria:

* Breast reconstruction using a TDAP or MSLD flap between January 1, 2018 and December 31, 2022
* Major
* Non opposition
* Women with social security number

Exclusion Criteria:

* Bilateral reconstruction
* Partial reconstruction
* Immediate reconstruction
* Prophylactic reconstruction
* Women who did'nt have a breast cancer
* Women who don't finish their reconstruction
* Women who don't want participate

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Women who underwent unilateral secondary total breast reconstruction using a TDAP or MSLD flap.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | 5 years
  patient satisfaction by using BREAST questionnaire (0 to 100, and 100 is the best score)

SECONDARY OUTCOMES:
Patient characteristics | 5 years
  Post-operative complications (number of hematoma, number of infection, number of seroma, number of flap lost), duration of the reconstruction (number of days), nature of additional interventions (number of lipofilling, symmetrization (yes or no), prothesis (yes or no))

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement